CLINICAL TRIAL: NCT01355133
Title: Transurethral Ultrasound-directed Injection of Autologous Myoblasts in Combination With Functional Electrical Stimulation in Patients With Intrinsic Urinary Sphincter Deficiency
Brief Title: Safety and Efficacy Study of Intrasphincteric Autologous Myoblast Injection to Treat Stress Urinary Incontinence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Innovacell Biotechnologie AG (Industry)
Responsible Party: Assoc. Prof. Adolf Lukanović, PhD, MD, Department of Gynecology, University Medical Center Ljubljana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Myoblast/ISD/EKS01; 2009-012389-30 (EudraCT Number)
Record Dates: First submitted 2011-05-12; First posted 2011-05-17 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Stress Urinary Incontinence
Keywords: Urinary incontinence; Myoblasts; Muscle derived cells; Stem cells
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Transurethral intrasphincteric autologous myoblast implantation — Patients undergo upper arm muscle biopsy to isolate and cultivate autologous myoblasts. Using the ultrasound-directed transurethral medical device, 15-18 aliquots (50 - 100 µl per depot) of the 2 ml myoblasts/media suspension are directly injected into the urethral rhabdosphincter at two different levels. The procedure is a single-dose injection of a cell count in range of 1x106 -5x107 cells, depending of the size/quality of the biopsy and quality of outgrowing cells in order to identify possible dose related effects. To possibly enhance cell integration following implantation, a course of transvaginal electrical stimulation is undertaken.

SUMMARY:
The purpose of this pilot clinical study is to determine if intrasphincteric autologous myoblast injections in combination with electrical stimulation are safe and effective in treating stress urinary incontinence, confirming the optimal dose and assessing tolerability of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Female outpatients, predominant clinical diagnosis of SUI
* Have discrete episodes of incontinence (that is, are dry between episodes and not continuously leaking urine, synchronous with increased intra-abdominal pressure from coughing, sneezing, exercising, etc.)
* Have a positive Fixed Bladder Volume Cough Stress Test (CST) result; and post void residual volume of <50 ml
* Report normal urinary diurnal (≤8/day) and nocturnal (≤2/night) frequency per micturition history
* Have had symptoms of SUI for a minimum of 3 months prior to study entry
* Can independently use toilet without difficulty
* If patients regularly use laxatives, stool softeners, or stool-bulking agents (for example, fibre supplements), the use of these products should remain constant during participation in the study.
* Competent to comprehend, sign, and date an Ethics Committee approved informed consent form before any study-specific procedure is performed.
* Are women of non-childbearing potential by reason of hysterectomy, other surgery, or natural menopause, or are women of childbearing potential who test negative for pregnancy at the time of enrolment based on a urine pregnancy test and agree to use a medically accepted means of contraception (for example, intrauterine device [IUD], oral or injectable contraceptives, implant, barrier device, sterilization, abstinence, or sex with a vasectomized male partner) for the duration of the study. Women using oral contraceptives or hormone replacement therapy must have a stable dose and regimen for greater than or equal to 3 months prior to entry into the study.

Exclusion Criteria:

* Previous diagnosis of any of the following conditions, disorders, or diseases of the urinary tract:

  * Greater than Stage I Anterior (cystocoele), Apical (uteri), or Posterior (rectocoele) Compartment Prolepses as per the POP-Q)
  * Ureteric bladder, urethral or rectal fistula
  * Uncorrected congenital abnormality leading to urinary incontinence
  * Interstitial cystitis
  * Urinary urgency that results in leakage (as a predominant symptom)
  * Adult enuresis
  * Urodynamically proven:
* detrusor instability
* sensory urgency defined as first sensation of bladder fill (urge to void) of <100 ml; bladder capacity of <300 ml
* voiding difficulty
* Have no sensation at any time during the simple filling cystometry procedure
* Unstable systemic disease including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months before enrollment
* Have a symptomatic urinary tract infection (UTI); or have a history of four or more urinary tract infections in the preceding year.
* Have prolonged menstruation (>14 days per month).
* Have history of (or currently have) urogenital cancer.
* Suffer from severe constipation defined as less than one bowel movement per week
* Are pregnant, <12 months postpartum or are lactating
* Have had any major inpatient surgery within 3 months prior to study entry
* Known infection with human immunodeficiency virus (HIV)
* Known active infection with Hepatitis B virus, Hepatitis C virus or Lues.
* Any organic or psychiatric disorder that, in the opinion of the investigator, might prevent the subject from completing the study or interfere with the interpretation of the study results.
* Have had any anti-incontinence or prolapse surgery, including the following:

  * Anterior Repair
  * Needle Suspension such as Raz; Pereyra; Stamey; Gittes; and Muzsnai procedures
  * Retropubic Procedures: such as Marshall, Marchetti & Krantz; and Burch procedures
  * Sling Procedure
  * Collagen Injections
  * Artificial Sphincter.
* Use any of the following:

  * Any anti-incontinence device (for example, Reliance, Minigard, or FemAssist) including tampons used to prevent incontinence during participation in the study
  * Vaginal pessaries for prolapse or incontinence
  * Any nonpharmacologic intervention for incontinence or prolapse (for example, electro stimulation, vaginal cones, or any such device) within the 3 months prior to study entry.
* Current use of any of the following drugs: antidepressants, duloxetine, monoamine oxidase inhibitors or other, clonidine, alpha-methyl-DOPA, beta-blockers, guanethidine, reserpine, pentosan polysulfate, or alpha-receptor antagonists/agonists (chronic use).
* Current use of any medications for the treatment of urinary incontinence.
* Are on a medication regimen including estrogens, anti-estrogens, or diuretics where dose and/or frequency has not been stable for at least the past 12 weeks, or is anticipated to change during the course of the study.
* ≤ 30 days since receiving an investigational medicinal product or device in another clinical trial. Current enrollment in another clinical trial is not permitted.
* Allergy/ intolerance of at least one of the active ingredients or excipients of the investigational products, e.g. bovine protein, gentamycin
* Have any abuse disorder within the 5 years prior to study entry; e.g. patients who report regular consumption of >21 alcoholic drinks per week (an average of 3 drinks per day)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Incontinence episode frequency (IEF) | 6 months post-implantation
  The median percent change from baseline in IEF using the 3-day bladder diary analysis
Change from baseline in Quality of Life (I-QOL) total score | 6 months post-implantation
  Mean improvement from baseline for the Incontinence Quality of Life (I-QOL) total score
Change from baseline in the Incontinence score | 6 months post-implantation

SECONDARY OUTCOMES:
Time to onset of response | Up to 6 months post-implantation (based on recordings at baseline, at implantation, at 6 weeks, 3 months and 6 months post-impalntation)
  Time to onset of response; time to maximum response; maintenance of response observed through changes in Incontinence episode frequency(IEF), Visual analog scale of the degree of suffering (VAS), Modified patient global impression of improvement(PGI-I*), fixed bladder stress test and I-QOL.
Change from baseline in Fixed bladder stress test outcome | Baseline, 6 months postimplantation.
Rate for subsequent incontinence surgery | 6 months post-implantation
Change from baseline in Urodynamic evaluation | 6 months post-implantation
  Cystometry, urethral pressure profile (UPP), 1-hour pad-test.
Safety | Up to 6 months post-implantation
  Number of adverse events, patholgical lab values, vital signs and weight recordings. Number of immediate and delayed complications of cell injection, including surgical injury, scars, urinary tract infection, inflammation, pelvic pain, prolonged urinary retention, voiding dysfunction, de novo urge incontinence, hematuria, hyperplasia or tumours.
  Any clinically significant findings based on physical examination, standard haematology, clinical chemistry and urinalysis profiles, Electrocardiogram (ECG), Blood Pressure (BP), pulse rate and adverse events recordings.
Change from baseline in Urinary incontinence semiquantitative (UIS) | 6 months post-implantation
  Amount of leaked urine measured semiqantitative from a 3-day bladder diary.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ljubljana, Dept. of Gynecology, Ljubljana, Slovenia

REFERENCES:
- [Derived] Blaganje M, Lukanovic A. Intrasphincteric autologous myoblast injections with electrical stimulation for stress urinary incontinence. Int J Gynaecol Obstet. 2012 May;117(2):164-7. doi: 10.1016/j.ijgo.2011.11.029. Epub 2012 Feb 18. PMID 22342057